CLINICAL TRIAL: NCT02362087
Title: A Multi-Centre Study to Investigate the Natural History of Taxane Acute Pain Syndrome (TAPS) in Patients Receiving Taxane Chemotherapy for Breast or Prostate Cancer
Brief Title: Taxane Acute Pain Syndrome (TAPS) in Patients Receiving Taxane Chemotherapy for Breast or Prostate Cancer
Acronym: TAPSOTT14-06
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20150011-01H
Record Dates: First submitted 2015-01-05; First posted 2015-02-12 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Acute Pain
Keywords: pain
MeSH Terms: conditions — Acute Pain; Pain | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma and buffy coat will be collected and archived tissure.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Quality of life and brief pain inventory — blood collection and quality of life questionnaires and a pain medication diary

SUMMARY:
The purpose of this study is to document what course of action physicians choose for their patients when they develop taxane acute pain syndrome (TAPS) and to identify patients at the greatest risk of TAPS by examining specific human genome markers such as single nucleotide polymorphisms (SNPs) and Copy Number Variations (CNVs) that may explain the genetic (hereditary) component.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with either invasive breast or prostate cancer (stage I-IV)
* Age ≥18 years
* ECOG performance status ≤2
* Scheduled to receive intravenous taxane-based chemotherapy for either adjuvant or metastatic disease
* Participants need to have ability to complete questionnaires by themselves or with assistance and have the ability to provide informed written consent

Exclusion Criteria:

* Concurrent use of any agents to try to prevent or treat neuropathy or TAPS, including gabapentin, glutamine, vitamin B6, and vitamin E.
* Pre-existing history of peripheral neuropathy greater than grade 1 NCI CTCAE version 4.0 from any cause (chemotherapy, diabetes, alcohol, toxin, hereditary, etc.) other medical conditions that would make study participation unreasonably hazardous
* Uncontrolled diabetes
* Medical or psychiatric illness that would interfere with patients' ability to complete the diary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Receiving Taxane Chemotherapy for Breast or Prostate Cancer
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The incidence of TAPS | Every 21 days over 12 weeks
  Participant will be asked prior to each taxane chemotherapy if they experienced TAPS and complete quality of life questionnaires

SECONDARY OUTCOMES:
The intervention used to reduced TAPS severity | Every 21 days over 12 weeks
  The intervention used to reduced TAPS severity including
  1. Analgesia - pain medication diary
  2. Exercise
  3. other
The TAPS associated treatment modification | Every 21 days over 12 weeks
  The TAPS associated treatment modification
  1. Taxane dose reduction
  2. Chemotherapy treatment delay
  3. Taxane discontinuation
  i. No further treatment pursued ii. Or Switch to non-taxane chemotherapy due to taxane toxicity
Collection of whole blood and archived tissue for future SNP analysis | At baseline and at one month from the end of Taxane chemotherapy
  Profiling of SNPs will aid to understand the genetic basis for TAPS and outcomes. We will also collect serum and plasma for profiling serum metabolites, drug metabolites and correlate with genotypes (SNPs)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Fernandes, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- Ricardo Fernandes, Ottawa, Ontario, Canada